CLINICAL TRIAL: NCT06327672
Title: INOCA Spanish National Registry: ESP-INOCA
Brief Title: INOCA Spanish National Registry
Acronym: ESP-INOCA
Status: Recruiting | Type: Observational
Sponsor: Eva Rumiz González (Other)
Collaborators: Hospital San Carlos, Madrid (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Hospital Universitario Virgen de la Arrixaca (Other); University Hospital Gregorio Marañón (Other); Hospital Clínico Universitario de Valladolid (Other); Hospital Universitario Puerta del Mar (Other); Hospital Universitari de Bellvitge (Other); Hospital Universitario La Fe (Other); Hospital Clínico Universitario de Valencia (Other); Hospital Universitario La Paz (Other); Hospital General Universitario de Alicante (Other); Complejo Hospitalario Universitario de Huelva (Other); Hospital General Universitario de Castellón (Other); Hospital de Manises (Other); Hospital Clinic of Barcelona (Other); Hospital Miguel Servet (Other); Hospital Clínico Universitario Lozano Blesa (Other); Hospital Donostia (Other); Hospital General Universitario Elche (Other); Hospital Universitario Virgen del Rocio (Unknown); Hospital de la Ribera (Other); Hospital de la Santa creu i Sant Pau - Barcelona (Other); Hospital Virgen de la Salud (Other); Hospital Universitario San Juan de Alicante (Other); Hospital Universitario de Torrevieja (Unknown); University Hospital of the Nuestra Señora de Candelaria (Other); Hospital de Basurto (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Universitario Fundación Jiménez Díaz (Other); Puerta de Hierro University Hospital (Other); Hospital Universitario 12 de Octubre (Other); University of Salamanca (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospital Clinico Universitario de Santiago (Other); Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Sponsor-Investigator, Eva Rumiz González, Principal Investigator, Hospital General Universitario de Valencia
Organization: Hospital General Universitario de Valencia (Other)
Other Study IDs: 162023
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Non-Obstructive Coronary Atherosclerosis; Ischemia; Coronary Disease
Keywords: Microvascular dysfunction; Endothelial dysfunction; Myocardial ischemia
MeSH Terms: conditions — Ischemia; Coronary Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronary atherosclerosis is the most common cause of ischaemic heart disease. About 40-50% of patients with symptoms and documented ischaemia on non-invasive tests do not show obstructive coronary artery disease on coronary angiography. This cause of ischaemic heart disease called INOCA (Ischemic Non-Obstructive Coronary Artery), far from having a benign prognosis, is associated with an increase in major adverse cardiac events (MACE) as well as increased functional limitation. The current European Society of Cardiology clinical practice guidelines for the management of chronic coronary syndrome establish for the first time a IIa recommendation for the invasive analysis of coronary flow reserve (CFR) and microvascular resistance index (MRI) in symptomatic patients with INOCA. The acetylcholine (Ach) test, based on intracoronary (ic) administration, is established as indication IIb for the assessment of micro or macrovascular vasospasm in patients with suspected vasospastic angina (VSA) (4). A national multicentre registry would allow us to determine the prevalence of INOCA and its different endotypes in our setting.

DETAILED DESCRIPTION:
Multicentre, observational, longitudinal, prospective study on INOCA patients undergoing invasive coronary function testing.

Microvascular angina (MVA) is defined according to the standardized diagnostic criteria of COVADIS (Coronary Vasomotion Disorders International Study Group): symptoms of myocardial ischaemia, unobstructed coronary arteries and demonstrated coronary microvascular dysfunction (CFR < 2 and/or IMR >25), or microvascular spasm on Ach test. Diagnosis of coronary microvascular spasm requires provocation and reproduction of symptoms, ischaemic EKG changes, in the absence of epicardial spasm during ACh testing. The diagnosis of VSA requires that 3 conditions are met during ACh testing: 1) clinically significant epicardial vasoconstriction (≥90%); 2) reproduction of chest pain; and 3) ischaemic EKG changes.

Definition of adverse events: Myocardial infarction (MI) will be defined according to the fourth universal definition and subclassified according to type. Ischaemia revascularization will be defined as all percutaneous coronary intervention (PCI) or Coronary Artery Bypass Grafting (CABG) occurring after the baseline procedure and justified by recurrent symptoms or objective evidence of significant ischaemia on non-invasive stress tests. Heart failure will be defined as a hospital admission > 24 hours with any of the following symptoms and signs: worsening dyspnea, fatigue, fluid overload, pulmonary oedema, elevated venous pressure and need for intravenous diuretics or inotropics. Visits to the emergency department for chest pain will be considered to be those in which there is suspicion of a coronary cause.

All events will be identified and quantified from patient records, including inpatient ward admissions and emergency department visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years.
* Anginal symptoms.
* Anginal equivalent with positive myocardial ischaemia test.
* Absence of obstructive coronary artery disease (diameter stenosis <50% or >50% with a FFR>0.80).
* Patients undergoing invasive coronary function test.
* Signed informed consent.

Exclusion Criteria:

* Failure to meet inclusion criteria.
* Patients with moderate-severe valvular heart disease.
* Patients with structural heart disease.
* Elevation of markers of myocardial necrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with angina and no obstructive coronary artery disease on coronary angiography, as well as those with angina equivalent symptoms and ischaemia on non-invasive tests (exercise stress test, cardiac magnetic resonance imaging, stress echocardiography, SPECT) in the absence of obstructive coronary artery disease, will be prospectively included. They must have undergone an invasive coronary function test. The absence of obstructive coronary artery disease will be defined as the presence of stenosis with a diameter <50% or >/= 50% and a negative functional test.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-24 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of INOCA endotypes. | 12 months
  To determine the prevalence of the different INOCA endotypes in our setting through a nationwide registry.

SECONDARY OUTCOMES:
Incidence of combined event: death from all causes, acute myocardial infarction, readmission for heart failure and consultation for chest pain in the emergency department. | 24 months
  To determine the long-term prognosis of the different INOCA subtypes, through analysis of the combined event: death from all causes, acute myocardial infarction, readmission for heart failure and consultation for chest pain in the emergency department.
Targeted pharmacological treatment | 24 months
  To determine the impact of targeted pharmacological treatment in INOCA patients.
Prognostic markers. | 24
  To identify prognostic markers.
INOCA and risk of heart failure with preserved ejection fraction. | 24 months
  To evaluate the association between INOCA patients and the development of heart failure with preserved ejection fraction.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Virgen de Arrixaca, Murcia
  - Hospital General Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Rumiz E, Rivero F, Perez A, Nau G, Romero M, Solana S, Jurado A, Fuertes G, Pardo A, Gutierrez-Barrios A, Casanova J, Oteo JF, Frutos A, Salvatella N, Cardenal R, Sabatel F, Cortes C, Valero E, Rodriguez R, Gutierrez E, Lopez-Palop R, Escaned J. ESP-INOCA: Rationale and design of a national multicentre registry for prognostic stratification in patients with suspected myocardial ischaemia and non-obstructive coronary arteries. Int J Cardiol. 2026 Jan 1;442:133845. doi: 10.1016/j.ijcard.2025.133845. Epub 2025 Aug 29. PMID 40886802